CLINICAL TRIAL: NCT04499768
Title: A Longitudinal Study of Choroidal Changes Assessed With Swept-source Optical Coherence Tomography After Cataract Surgery in Eyes With Diabetic Retinopathy
Brief Title: A Longitudinal Study of Choroidal Changes After Cataract Surgery in Eyes With Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xi Shen, chief physician, Ruijin Hospital
Other Study IDs: 2018ZY14
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Optical Coherence Tomography; Diabetic Retinopathy; Choroid
Keywords: Diabetic choroidopathy; Diabetic retinopathy; choroidal vascularity index; choroidal thickness
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: the age-related cataract patients
- DR group: the cataract patients with mild/moderate NPDR

SUMMARY:
To determine the influence of phacoemulsification on choroidal vasculature in patients with diabetic retinopathy (DR) undergoing cataract surgery

DETAILED DESCRIPTION:
To determine the influence of phacoemulsification on choroidal vasculature in patients with diabetic retinopathy (DR) undergoing cataract surgery through the follow-up of choroidal thickness (CT) and choroidal vascularity index (CVI) using swept-source optical coherence tomography (SS-OCT) system.

ELIGIBILITY:
Inclusion Criteria:

* aged⩾40years; intraocular pressure (IOP) < 21 mm Hg in both eyes, spherical refractive error<6 diopters spherical equivalent.

Exclusion Criteria:

* previous retinal surgery, glaucoma, uveitis, age-related macular degeneration, arterial or vein occlusions, macular hole, or other ocular diseases that could interfere the CT and/or CVI measurement, severe systemic diseases, such as uncontrolled hypertension, obstructive sleep apnea, etc.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 23 eyes of 23 cataract patients with mild/moderate NPDR without DME, and 23 age-matched non-diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
CVI at baseline | CVI was assessed at baseline(within 1 week before surgery)
  choroidal vascularity index(CVI) was defined as the proportion of vascular area to total circumscribed area.
CVI at 1 week postoperatively | CVI was assessed 1 week after surgery.
  choroidal vascularity index (CVI) was defined as the proportion of vascular area to total circumscribed area.
CVI at 1 month postoperatively | CVI was assessed 1 month after surgery.
  choroidal vascularity index (CVI) was defined as the proportion of vascular area to total circumscribed area.
CVI at 3 months postoperatively | CVI was assessed 3 months after surgery.
  choroidal vascularity index (CVI)was defined as the proportion of vascular area to total circumscribed area.
CT at baseline | CT was assessed at baseline and 1 week, 1 month, 3 month after surgery.
  Choroid thickness (CT) was the thickness of the choroidal layer; CT values were obtained with the built-in software of the SS-OCT device.
CT at 1 week postoperatively | CT was assessed at 1 week after surgery.
  Choroid thickness (CT) was the thickness of the choroidal layer; CT values were obtained with the built-in software of the SS-OCT device.
CT at 1 month postoperatively | CT was assessed at 1 month after surgery.
  Choroid thickness (CT) was the thickness of the choroidal layer; CT values were obtained with the built-in software of the SS-OCT device.
CT at 3 months postoperatively | CT was assessed at 3 months after surgery.
  Choroid thickness (CT) was the thickness of the choroidal layer, CT values were obtained with the built-in software of the SS-OCT device.
VD at baseline | VD of the choriocapillaris was assessed at baseline.
  VD of the choriocapillaris was the vessel density of the choriocapillaris in the choroid.
VD at 1 week postoperatively | VD of the choriocapillaris was assessed 1 week after surgery.
  VD of the choriocapillaris was the vessel density of the choriocapillaris in the choroid.
VD at 1 month postoperatively | VD of the choriocapillaris was assessed 1 month after surgery.
  VD of the choriocapillaris was the vessel density of the choriocapillaris in the choroid.
VD at 3 months postoperatively | VD of the choriocapillaris was assessed 3 months after surgery.
  VD of the choriocapillaris was the vessel density of the choriocapillaris in the choroid

SECONDARY OUTCOMES:
IOP at baseline | IOP was assessed at baseline and 1 week, 1 month, 3 month after surgery.
  IOP was the value of intraocular pressure.
IOP at 1 week postoperatively | IOP was assessed 1 week after surgery.
  IOP was the value of intraocular pressure .
IOP at 1 month postoperatively | IOP was assessed 1 month after surgery.
  IOP was the value of intraocular pressure.
IOP at 3 months postoperatively | IOP was assessed 3 months after surgery.
  IOP was the value of intraocular pressure .
BCVA at baseline | BCVA was assessed at baseline .
  BCVA was the best corrected visual acuity.
BCVA at 3 months postoperatively | BCVA was assessed 3 months after surgery.
  BCVA was the best corrected visual acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Shen, PhD, Study Director — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Yao H, Gao S, Liu X, Zhou Y, Cheng Y, Shen X. Choroidal Structural Changes Assessed with Swept-Source Optical Coherence Tomography after Cataract Surgery in Eyes with Diabetic Retinopathy. J Ophthalmol. 2020 Oct 29;2020:5839837. doi: 10.1155/2020/5839837. eCollection 2020. PMID 33178452